CLINICAL TRIAL: NCT03651453
Title: Developing and Testing the Effect of a Patient-Centered HIV Prevention Decision Aid on PrEP Uptake for Women With Substance Use in Treatment Settings
Brief Title: OPTIONS: A Patient-Centered HIV Prevention Decision Aid for PrEP Uptake for Women With Substance Use in Treatment Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000021561
Record Dates: First submitted 2018-08-01; First posted 2018-08-29 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: HIV Infections; Substance Abuse
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders | interventions — Decision Support Techniques; Standard of Care; Therapeutics

STUDY DESIGN:
Intervention Model Description: A controlled un-blinded pilot study.
Masking Description: A controlled un-blinded pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Participants will receive standard information about harm reduction as available at the drug treatment centers.
  Interventions: Behavioral: Standard care
- Decision aid (Experimental): Participants in this arm will receive the adapted decision aid for PrEP.
  Interventions: Behavioral: Decision aid

INTERVENTIONS:
Behavioral: Decision aid — Participants in the experimental arm will receive the PrEP decision aid.
  Other Names: PrEP decision aid
  Arms: Decision aid
Behavioral: Standard care — Standard harm reduction information
  Other Names: treatment as usual
  Arms: Standard Care

SUMMARY:
To develop and test the effect of a patient-centered HIV prevention decision aid on HIV pre-exposure prophylaxis (PrEP) uptake among women with substance use disorders (SUD) in treatment.

DETAILED DESCRIPTION:
To test the effect of the informed decision aid intervention on PrEP uptake among women with substance use disorders in treatment. Investigators hypothesize that compared to those receiving standard harm reduction information, women receiving the decision aid will have a significant increase in PrEP uptake at 6 and 12 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Self- identification as female (i.e., cis- or trans- women), age ≥18, HIV negative status (confirmed with APT date from rapid testing procedures), and entering or receiving treatment at our partnering site, the APT Foundation, Inc. (a drug treatment center).

Exclusion Criteria:

* Women on PrEP at baseline, unable or unwilling to provide informed consent, threatening to staff, pregnant, or experiencing symptoms of physiological withdrawal that interfere with ability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — cis- or trans- female eligible
Enrollment: 164 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
PrEP Uptake | 12 months
  PrEP uptake is measured by attending an appointment with a provider for the purposes of starting PrEP.

SECONDARY OUTCOMES:
PrEP Adherence by Self Report | 12 months
  Adherence to PrEP is measured by pill count
PrEP Adherence by Pharmacy Refill | 12 months
  Adherence to PrEP is measured by pharmacy refill data
Changes in PrEP receptiveness | 12 months
  Receptiveness to PrEP (pre- and post- decision aid) is measured on a receptiveness scale (Likert 1-5)
Changes in HIV risk behaviors | 12 months
  Changes in HIV risk is measured by a modified risk assessment form from NIDA

CONTACTS AND LOCATIONS:
Overall Officials: Jaimie P Meyer, MD, Principal Investigator — Yale University
Locations (1):
- Yale AIDS Program, New Haven, Connecticut, United States